CLINICAL TRIAL: NCT06275438
Title: Comparison of Oxytocin Receptor Immunoreactivity in Placentas Obtained From Women Having Cesarean and Natural Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Şevin Akgün, research assistant, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 81829502.903/39
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy Mothers Who Have Had Both Vaginal and Cesarean Deliveries
Keywords: Cesarean Section, Decidua, Midwife, Oxytocin Receptor, Placenta

STUDY DESIGN:
Intervention Model Description: "Our study was conducted on the placentas of 40 women admitted to the obstetrics clinics of Kars Harakani State Hospital and Kafkas University Training and Research Hospital, after obtaining necessary permissions. Out of 40 placentas, 5 were excluded due to blood incompatibility, 2 were excluded due to subsequent diagnosis of chronic conditions (thyroid disorder, Behçet's disease), and 1 was excluded due to the presence of an accessory placenta, resulting in a total of 32 placentas included in the study. Among these, 16 were from women who had undergone normal vaginal delivery (control group), and 16 were from women who had undergone cesarean section (case group). Tissue samples obtained from the placentas were subjected to histological and immunohistochemical methods to obtain various findings
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Active Comparator): The group consists of mothers who meet the inclusion criteria specified in the study, have an 8cm dilation at term, and undergo cesarean section delivery.
  Interventions: Other: The delivery being performed via cesarean section surgery rather than natural childbirth
- control group (No Intervention): The group comprises healthy mothers who meet the inclusion criteria specified in the study, have an 8cm dilation at term, and give birth vaginally.

INTERVENTIONS:
Other: The delivery being performed via cesarean section surgery rather than natural childbirth — At Kars Harakani State Hospital and Kafkas University, 16 placentas were collected, with 8 obtained from induced deliveries and 8 from spontaneous deliveries, between 09:00-21:00. Nulliparity and multiparity were not distinguished among the expectant mothers. Placentas were obtained hours before delivery from mothers admitted to the gynecology service, whose eligibility was determined based on exclusion criteria, after obtaining signed informed consent forms, with assurances given that no interventional procedures would be performed on the mother or the baby. The method of cesarean section (spinal or general anesthesia) in the case group was recorded, ensuring that the anesthetic agents used contained the same active ingredients. Placentas from births involving different anesthetic drugs were not included in the study, aiming to standardize the procedure.
  Arms: experimental group

SUMMARY:
Our study examines the effects of oxytocin hormone receptors. mechanisms of placental tissue cells and therefore intrauterine development. It was conducted to investigate the effects on newborn babies apgar score, fontanel openings, birth weights, etc. By collecting data, normal and They were compared between cesarean births by statistical analysis. normal in this regard Based on the hypothesis that there is a difference between labor and cesarean delivery, this study has been made.OXTR primary antibody was used for immunohistochemical examination. There was no significant difference between the groups in terms of histological examination. In the study, it was found that OXTR immunoreactivity was strong in decidual cells and stromal cells in villi. A stronger OXTR immunoreactivity was detected in villous stroma of placenta of the natural birth group compared to the cesarean birth group. Reaction was not observed in syncytotrophoblast cells and syncytial nodes in both groups, but strong immunoreaction was observed fetal endothelial cells and fetal capillaries in both groups.

DETAILED DESCRIPTION:
The aim of this study was to compare oxytocin receptor (OXTR) immunoreactivity in placentas obtained from women having cesarean and natural birth. The study samples consisted of placentas of 32 mothers who had 16 natural birth (control) and 16 cesarean (case) birth in Kars Harakani State Hospital and Kafkas University Health Research and Application Hospital. At the beginning of the study, 40 placentas obtained in total, 5 were not included in the study due to mismatched blood, 2 were not included in the study after the chronic disease (thyroid, Behçet's disease) detected, and 1 was not included in the study due to the presence of accessory placenta. The means of binary variables were determined by applying the Independent Two-Sample T-Test. Pearson Correlation analysis was used to examine the relationship between the variables. Periodic acid-Schiff staining, H&E and Triple staining techniques were applied to tissue samples obtained from placentas for histological examination. OXTR primary antibody was used for immunohistochemical examination. There was no significant difference between the groups in terms of histological examination. In the study, it was found that OXTR immunoreactivity was strong in decidual cells and stromal cells in villi. A stronger OXTR immunoreactivity was detected in villous stroma of placenta of the natural birth group compared to the cesarean birth group. Reaction was not observed in syncytotrophoblast cells and syncytial nodes in both groups, but strong immunoreaction was observed fetal endothelial cells and fetal capillaries in both groups. As a result, it is thought that the placenta pathology should be made routine for every birth because it gives information about the offspring.

ELIGIBILITY:
Inclusion Criteria:

Mothers with a body mass index within this range:18kg/m2≥Body Mass Index (BMI)≤35kg/m2 Healthy mothers who have had both vaginal and cesarean deliveries Mothers aged over 18 and under 35 years old

Exclusion Criteria:

* Chronic diseases Gynecological disorders Intrauterine growth restriction Placental anomalies Forensic cases of pregnancy Premature births Eclampsia-Preeclampsia Multiple pregnancies Body Mass Index (BMI) ≥35kg/m2 Body Mass Index (BMI) ≤18kg/m2 Experience of trauma during pregnancy Non-cesarean surgical interventions during pregnancy Severe infections

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy mothers who have had vaginal and cesarean deliveries
Enrollment: 32 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Oksitosin Receptor Immunoreactivity | 2 weeks
  After subjecting the placenta samples to various biochemical tests and staining procedures, they were prepared appropriately and evaluated for oxytocin receptor activity after being incubated for 24 hours.

SECONDARY OUTCOMES:
Pearson correlation analysis | 1 months
  The collected data included variables such as maternal age, body mass index (BMI), number of abortions, number of abortions, age at first pregnancy, number of live children, date of last menstrual period, and various newborn parameters such as gender, weight, head circumference, length, 1st and 5th minute Apgar scores, anterior-posterior fontanelle opening, placental thickness, weight, major-minor diameter, and total cord length.
  For the statistical analysis of the collected data, version 20.0 of the SPSS program was utilized. Independent Samples T-Test was applied to compare the means of binary variables and their differences at a significance level of 5%. Pearson correlation analysis was employed to examine the relationships between variables.

CONTACTS AND LOCATIONS:
Overall Officials: Seyit Ali Bingöl, associate professor dr., Study Director — Kafkas University Faculty of Medicine; SEVİN Polat, resarch assistant, Study Chair — Kafkas University Faculty Of Health Sciences
Locations (1):
- Kafkas Universty, Kars, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The participants were explicitly informed in the voluntary consent form that their information and the data obtained from the study would not be used for any other study and would not be shared with a third party. Participation in the study was contingent upon the condition that their confidentiality would be protected.

REFERENCES:
- [Result] Aydogan A, Bingol SA. Examination of the immunohistochemical localization and gene expression by RT-PCR of the oxytocin receptor in diabetic and non-diabetic mouse testis. Iran J Basic Med Sci. 2018 Jul;21(7):695-700. doi: 10.22038/IJBMS.2018.28069.6820. PMID 30140408
- [Result] Szukiewicz D, Bilska A, Mittal TK, Stangret A, Wejman J, Szewczyk G, Pyzlak M, Zamlynski J. Myometrial contractility influences oxytocin receptor (OXTR) expression in term trophoblast cells obtained from the maternal surface of the human placenta. BMC Pregnancy Childbirth. 2015 Sep 16;15:220. doi: 10.1186/s12884-015-0656-3. PMID 26377392
- [Result] Barker DJ, Thornburg KL, Osmond C, Kajantie E, Eriksson JG. The surface area of the placenta and hypertension in the offspring in later life. Int J Dev Biol. 2010;54(2-3):525-30. doi: 10.1387/ijdb.082760db. PMID 19876839
- [Result] Buisman-Pijlman FT, Sumracki NM, Gordon JJ, Hull PR, Carter CS, Tops M. Individual differences underlying susceptibility to addiction: Role for the endogenous oxytocin system. Pharmacol Biochem Behav. 2014 Apr;119:22-38. doi: 10.1016/j.pbb.2013.09.005. Epub 2013 Sep 18. PMID 24056025
- [Result] Alwasel SH, Harrath A, Aljarallah JS, Abotalib Z, Osmond C, Al Omar SY, Khaled I, Barker DJ. Intergenerational effects of in utero exposure to Ramadan in Tunisia. Am J Hum Biol. 2013 May-Jun;25(3):341-3. doi: 10.1002/ajhb.22374. Epub 2013 Feb 21. PMID 23436278
- [Result] Eriksson JG, Gelow J, Thornburg KL, Osmond C, Laakso M, Uusitupa M, Lindi V, Kajantie E, Barker DJ. Long-term effects of placental growth on overweight and body composition. Int J Pediatr. 2012;2012:324185. doi: 10.1155/2012/324185. Epub 2012 Apr 18. PMID 22570665
- See also: Maternal blood and amnionic oxytocin receptor gene expression and serum oxytocin levels in preterm birth: a case control study — http://www.medrxiv.org/content/10.1101/2020.07.18.20155879v1